CLINICAL TRIAL: NCT06931548
Title: Ways of Retaining the Inframammary Fold in Implant-based Breast Surgery Using Polytetrafluoroethylene (PTFE) Mesh or Allogeneic Dura Mater Graft
Brief Title: Ways of Retaining the Inframammary Fold in Implant-based Breast Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Branch Office of "Hadassah Medical Ltd" (Other)
Collaborators: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREAST-ONE
Record Dates: First submitted 2025-04-06; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; In Situ Breast Cancer
Keywords: implant-based breast reconstruction; breast cancer; PTFE mesh
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polytetrafluoroethylene mesh (Experimental): Patients in this group will undergo one-stage breast reconstruction using an implant and polytetrafluoroethylene (PTFE) mesh after subcutaneous or skin-sparing mastectomy.
  Interventions: Procedure: Implant-based breast reconstruction using polytetrafluoroethylene mesh
- Allogeneic dura mater graft (Active Comparator): Patients in this group will undergo one-stage breast reconstruction using an implant and allogeneic dura mater graft after subcutaneous or skin-sparing mastectomy.
  Interventions: Procedure: Implant-based breast reconstruction using Allogeneic dura mater graft

INTERVENTIONS:
Procedure: Implant-based breast reconstruction using polytetrafluoroethylene mesh — Patients will undergo subcutaneous or skin-sparing mastectomy using the standard technique. Simultaneously, breast reconstruction will be performed using a breast implant. The lower pole of the implant and the inframammary fold will be additionally reinforced with polytetrafluoroethylene (PTFE) mesh. The lower edge of the mesh is sutured in the projection of the inframammary fold, and the upper edge is sutured to the pectoralis major muscle.
  Arms: Polytetrafluoroethylene mesh
Procedure: Implant-based breast reconstruction using Allogeneic dura mater graft — Patients will undergo subcutaneous or skin-sparing mastectomy using the standard technique. Simultaneously, breast reconstruction will be performed using a breast implant. The lower pole of the implant and the inframammary fold will be additionally reinforced with an allogeneic dura mater graft. The lower edge of the mesh is sutured in the projection of the inframammary fold, and the upper edge is sutured to the pectoralis major muscle.
  Arms: Allogeneic dura mater graft

SUMMARY:
There is currently no consensus on the "gold standard" for Implant-based Breast reconstruction. In the United States, more than half of all breast reconstructions are performed using acellular dermal matrix (ADM). However, based on the findings of literature and systematic reviews, it can be cautiously said that synthetic meshes cause fewer complications with comparable aesthetic results and low cost. In our study, we propose using polytetrafluoroethylene (PTFE) mesh in implant-based breast reconstruction. This material has previously proven itself in cardiovascular, maxillofacial and neurosurgery, hernioplasty and as a suture material. Allogeneic dura mater, which has demonstrated comparable results in breast reconstruction with the literature, will be used as a comparison. The purpose of this study is to evaluate the efficacy and safety of a porous, non-biodegradable, synthetic polytetrafluoroethylene mesh for implant-based breast reconstruction in patients diagnosed with breast cancer. An allogeneic dura mater technique will be used as a control.

Patients eligible for this study are classified according to the National Comprehensive Cancer Network (NCCN) guidelines as having stage 0-2 breast cancer.

The primary questions this study aims to answer are:

* What are the rates of major and minor complications associated with these techniques. Major complications will be defined as complications leading to reoperation.
* How effective are PTFE mesh and dura in maintaining the inframammary fold and implant projection after breast reconstruction?
* What is the patient satisfaction rate with the surgical results?

Patients will be randomly assigned to the study but will know which technique will be used in their particular case. Patients included in this study will undergo subcutaneous mastectomy or skin-sparing mastectomy using standard techniques with simultaneous implantation using PTFE mesh or allogeneic dura mater graft. In our opinion, the mesh and graft will stabilize the projections of the inframammary fold and breast implant.

After the surgery, all minor and major complications will be recorded for 6 months. For this, both physical examination and radiological diagnostic methods will be used, including breast ultrasound and MRI with contrast. Revision surgeries will be performed if necessary.

Projections of the inframammary fold and breast implant will also be measured in order to determine the effectiveness of the compared techniques.

Patients will be asked to complete the BREAST-Q Version 2.0© Reconstruction Module questionnaire to determine satisfaction with the surgical outcome.

The results of the study will help the professional community to determine the most effective method of Implant-based Breast reconstruction and will be published in peer-reviewed scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* White women;
* Breast cancer stage 0-II;
* Indications for breast reconstruction;
* Consent to participate in the study and photographic documentation.

Exclusion Criteria:

* Non-white women;
* Breast cancer stage III-IV;
* Tubular breast;
* Mental and cognitive health disorders;
* Failure to comply with recommendations in the postoperative period (premature physical activity, not wearing compression underwear, missing scheduled visits, refusal of photo documentation);
* Patient refusal to participate in the study at any stage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of major and minor complications | within 6 months from the date of surgery
  Major complications will be defined as complications that lead to revision surgery. These may include long-term seromas and hematomas, necrosis, infections that are not controlled by therapy or physical therapy. Also, displacement of the implant position by more than 2 cm.
  Minor complications will be defined as complications that do not require reoperation.

SECONDARY OUTCOMES:
Evaluation of changes in projections of the implant and inframammary fold | within 6 months from the date of surgery
  After the operation and after 6 months, the following distances will be measured:
  * from the jugular notch to the nipple;
  * from the middle of the clavicle to the nipple;
  * from the anterior midline to the nipple;
  * from the inframammary fold to the nipple.
  Calipers are used for measurements, distances are measured in the metric system. These measurements will allow you to assess the change in the position of the implant and, as a result, the shape of the breast. Changes in distances immediately after surgery and the same distances after 6 months by more than 1 cm (0.39 inches) will be considered a significant displacement of the implant.
Quality of life | within 6 months from the date of surgery
  After surgery and 6 months later, patients will be asked to complete the BREAST-Q Version 2.0© Reconstruction Module questionnaire:
  * "Physical well-being: chest";
  * "Sexual well-being";
  * "Psychosocial well-being";
  * "Satisfaction with breast".
  The BREAST-Q© is a rigorously developed patient-reported outcome (PRO) measure designed to evaluate outcomes among women undergoing different types of breast surgery. In this study, the "Reconstructive Module" of the questionnaire will be used.
  There is no overall or total BREAST-Q© score, only scores for each independent scale. All BREAST-Q© scales are transformed into scores that range from 0-100. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q© scales, a higher score means greater satisfaction or better QOL (depending on the scale).

CONTACTS AND LOCATIONS:
Overall Officials: Alla Kartasheva, PhD, Principal Investigator — The Branch of Hadassah Medical LTD
Locations (1):
- The Branch of Hadassah Medical LTD, Moscow, Skolkovo Innovation Center, Russia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in a publication will be formed into a single tabular data array and placed in cloud storage. Access to viewing this array will be provided upon request of researchers or scientific publications (through the corresponding author).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: The data obtained as a result of the study will be published in scientific journals in general form. Accordingly, we see no reason not to provide access to the original data - the data array. In case of interest in the array and any additional information, it will be necessary to contact the members of the research group - the co-authors of the publication. According to generally accepted rules, when publishing an article, the e-mail address of at least one of the co-authors is indicated. Thus, if necessary, interested parties can write to the co-authors directly to provide access.